CLINICAL TRIAL: NCT04149236
Title: A Qualitative Study of Cultural Perception of Health in Rural Guatemala
Acronym: deCiPHeRGap
Status: Withdrawn | Type: Observational
Why Stopped: Was halted during the COVID pandemic; study continuation plans discontinued as some investigators no longer associated with the University of Colorado.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1828
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Qualitative Research; Beliefs
Keywords: Culture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Investigators will be giving a survey to ~100 people in a rural community in Guatemala to discover beliefs and perspectives that the Participants have surrounding various aspects of healthcare. The Investigators aim to do this in order to be able to better serve the population in the community by discovering specific information about them from the Participants and how the Participants about different health practices. The Investigators will answer their research questions through the questionnaire that will allow participants to explain their viewpoints about a variety of medical topics.

DETAILED DESCRIPTION:
The design of this cross-sectional study is centered around a structured questionnaire of a mixed qualitative and quantitative nature that is composed primarily of yes/no or Likert scale responses. All questions are written with the intent that they may be understood by those participants without any formal education. The investigators will recruit participants that are currently using the services of the Trifinio clinic in rural Guatemala as these are likely to fit inclusion criteria and will be able to benefit from potential future services that will be directed by the findings of this questionnaire. For all participants, Likert scale questions will be used with a series of faces to help indicate meanings for the answers and to decrease possibility of misinterpretation. Participants will be recruited through non-probabilistic sampling and the use of snowball sampling. Screening of these participants for exclusion criteria will be performed before questionnaires are distributed. The questions of the questionnaire are designed to elicit information about certain beliefs or preferences related to healthcare in a structured manner that allows us to compare answers and determine trends, prevalence, and associations that are likely to exist among community members. Participation will be completely voluntary and informed consent will be obtained from each participant before they are given the questionnaire. For participants who are illiterate or would prefer to have the informed consent and questionnaire read aloud to them, this will be done by one of the CITI-trained investigators. Recorded data will only include questionnaire responses and will not include any identifying information. We will be using randomized numbers in order to refer to completed questionnaires, but these numbers will have no identifying aspects and will be used for the sole purpose of keeping track of the gathered data. The information gathered will be de-identified and stored and password-protected through REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Willing and able to participate in the questionnaire (if participant is illiterate, they will have the option to have each question and all responses read to them aloud by one of the trained researchers)
* Live in one of the communities within 50 km of the research site
* Those participants born in Guatemala

Exclusion Criteria:

* < 18 or >64 years old
* Decisionally challenged
* Refusal or inability to give consent
* Those born outside of Guatemala
* Those living in areas > 50 km from the research site

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of local rural Guatemalans that live within 50 km of the clinic site that wish to participate in completing a questionnaire to better inform the clinic of community needs, educational opportunities, and available resources.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of Gaps in Knowledge Surrounding Health Services | Day 1
  A survey with yes/no questions whether a participant is aware of health services available to them. Answers will be scored as 1 = Yes/Aware or 0=No/Not Aware.
Perceptions of Healthcare, as Determined by Agreeability of Statements | Day 1
  Likert scale responses will be shown to participants who will choose among 5 answers ranging from "Very Much So Disagree" to "Very Much So Agree". The answers chosen will be summed and put into percentages that each answer receives, demonstrating prevalence of those beliefs among the participants.

CONTACTS AND LOCATIONS:
Overall Officials: James L Martin, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No
The Investigators will de-identify participants and pool total data after questionnaire completion. The results of pooled data may be shared but individual participant data will not be.